CLINICAL TRIAL: NCT06978062
Title: An Open-label, Multi-centre, Phase 1b Safety and Feasibility Study for the Peri-operative Treatment of Resectable Gastroesophageal Cancer Using Bemarituzumab (BEMA) Plus Perioperative Treatment (NeoBEMA)
Brief Title: Peri-operative Treatment of Resectable Gastroesophageal Cancer Using Bemarituzumab (BEMA) Plus Perioperative Treatment
Acronym: NeoBEMA
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC 2385-GITCG
Record Dates: First submitted 2025-04-29; First posted 2025-05-18 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: GastroEsophageal Cancer
MeSH Terms: interventions — bemarituzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FLOT plus Bemarituzumab (Experimental): * FLOT will be administered every 2 weeks (Q2W). Docetaxel 50 mg/m2 is given as 1 hour infusion, followed by Oxaliplatin 85mg/m2 as a 2-hour infusion, leucovorin 200 mg/m2 over 2 hours and 5-FU 2600 mg/m2 as a 24 hour-infusion,
  * Bemarituzumab will be administered as IV infusion
  Interventions: Drug: Bemarituzumab; Drug: FLOT

INTERVENTIONS:
Drug: Bemarituzumab — • Bemarituzumab will be given as a IV infusion
Drug: FLOT — FLOT will be given as a IV infusion

SUMMARY:
This is an open-label,multi-centre, phase 1b safety and feasibility study aiming to assess the safey and feasibility of bemarituzumab plus chemiotherapy (FLOT) for the peri-operative treatment of resectable gastroesophageal cancer. Following this neo-adjuvant part, patients should undergo surgery. Following surgery, patients will receive FLOT chemotherapy in combination with bemarituzumab. Imaging will be performed every 3 months for the first 2 years and thereafter every 6 months as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Signed screening informed consent
* Age ≥ 18 years
* Availability of a diagnostic tumour sample for central evaluation (FFPE block or minimum 10 slides).
* Histologically proven, previously untreated, locally advanced, resectable gastric/GEJ adenocarcinoma cT2-cT4, N0, M0 or cTany, N+, M0. Note: if the results of the staging laparoscopy are pending at this stage it is acceptable to include the patients in this step, in the interest of patient time-to-treatment.
* Planned peri-operative treatment with FLOT chemotherapy and surgically assessed feasible R0 resection
* Centrally confirmed FGFR2b overexpression as defined by ≥10% tumour cells with 2+/3+ FGFR2b staining by immunohistochemistry (IHC)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Previously untreated, locally advanced, histologically confirmed, resectable gastric/GEJ adenocarcinoma cT2-cT4, N0, M0 or cTany, N+, M0 by radiological and surgical staging
* Adequate hematologic and organ function

Exclusion Criteria:

* Prior anticancer treatment for the disease under investigation
* History or evidence of systemic disease or ophthalmological disorders requiring chronic use of ophthalmologic corticosteroids
* Evidence of any ongoing ophthalmologic abnormalities or symptoms that are recent (within 4weeks) or actively progressing
* Unwillingness to avoid the use of contact lenses during study treatment and follow-up period of at least 100 days after end of treatment.
* Evidence of, or recent (within 6 months) history of, corneal defects, corneal ulcerations, keratitis, or keratoconus, history of corneal transplant, or other known abnormalities of the cornea that may pose an increased risk of developing a corneal ulcer. Recent (within 6 months) corneal surgery or ophthalmologic laser treatment
* History of solid organ transplantation
* History of interstitial lung disease
* Active autoimmune disease that has required systemic treatment (except replacement therapy) within the past 2 years or any other diseases requiring immunosuppressive therapy while on study
* Patients on immunosuppressive therapy or having immune system disorders, including auto-immune diseases. Concurrent steroid use of not more than an equivalent of 10 mg/day prednisolone is allowed. Inhaled, intranasal, intraocular, and/or joint injections of corticosteroids are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2028-09-11 (Estimated); Study Completion 2029-09-28 (Estimated)

PRIMARY OUTCOMES:
Completion rate of neoadjuvant treatment followed by surgery without serious anastomotic leakage, defined as the percentage of patients who completed the treatment without grade 2 or more anastomotic leakage as per Clavien-Dindo Classification | 2.3 years from first patient in
  Patients will be considered to have successfully completed the neo-adjuvant treatment if they complete the 4 cycles of FLOT plus Bemarituzumab. Additionally, anastomotic leakage will be reported as post-surgery complication following the modified Clavien-Dindo Classification

SECONDARY OUTCOMES:
Major pathological response | 3.6 years from first patients in
  Major pathological response rate will be computed as the percentage of patients who had major tumour regression (< 10% vital residual tumour cells) after neoadjuvant treatment.
Pathological complete response | 3.6 years from first patients in
Progression free survival (PFS) | 3.6 years from first patients in
  Progression-free survival is defined as the time interval from enrolment to the first event of progression/recurrence
Overall survival (OS) | 3.6 years from first patients in
  Overall survival will be computed from the date of enrolment to the date of death
Treatment-emergent adverse events | 3.6 years from first patients in
R0 resection | 3.6 years from first patients in
Completion rate of neoadjuvant and adjuvant therapy | 3.6 years from first patients in
Postoperative complications according to CLAVIEN DINDO classification | 3.6 years from first patients in
30 and 90 day-mortality after surgery | 1.7 years from first patients in

CONTACTS AND LOCATIONS:
Overall Officials: Markus Moehler, Principal Investigator — University Medical Center Mainz; Elizabeth Smyth, Principal Investigator — University of Oxford; Maike Collienne, Principal Investigator — University Medical Center Mannheim